CLINICAL TRIAL: NCT04573998
Title: Study on the Mechanism of lcn2 in Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shen Qu (Other)
Responsible Party: Sponsor-Investigator, Shen Qu, Principal Investigator, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: LCN2
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Endocrine
Keywords: obesity; lcn2
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: LSG — bariatric surgery

SUMMARY:
Obesity is now becoming a worldwide serious problem. Obesity is associated with a spectrum of severe diseases, including diabetes, cardiovascular diseases, and cancers. Lipocalin 2 (LCN2), also known as neutrophil gelatinase associated lipocalin (NGAL), is a member of the lipocalin family. Due to its upregulated expression in infection, LCN2 is originally considered to be a key regulator of immune response. Subsequent investigations revealed that LCN2 is expressed in many tissues and is related to a variety of diseases, including obesity. LCN2 was reported to be increased in obesity individuals. Thus, the investigators decide to investigate the relationship between LCN2 and obesity.

ELIGIBILITY:
Inclusion Criteria:

1) age ranged from 16-65 years old, 2) BMI over 37.5kg/m2, or BMI over 32.5kg/m2 with diabetes which meets the recommended cut off bariatric surgery of the Guidelines for surgical treatment of obesity accompanied with or without type 2 diabetes in China.

Exclusion Criteria:

1) secondary cause of obesity such as hypothalamic obesity, Cushing syndrome, and hypophysis dysfunction, etc.,2)pregnancy or location, 3) contraindications for laparoscopic surgery, such as gastrointestinal diseases of intra-abdominal infection, adhesion, etc., 4) severe heart, liver and kidney dysfunction, 5) organic and systemic diseases intolerant of surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 500 Patients from Shanghai Tenth People's Hospital were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
LCN2 level | 2019-2024
  Lipocalin 2 level
meet the criteria of metabolism in the 2017 Chinese guideline | 2019-2024
  Abdominal obesity (or central obesity), male abdominal circumference ≥90cm, female abdominal circumference ≥85cm;

SECONDARY OUTCOMES:
FBG | 2019-2024
  patients with fasting blood glucose 6.1mmol/l or more
PBG | 2019-2024
  patients with 2 hour blood glucose 7.8mmol/l or more

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Dr., Study Chair — Shanghai 10th People's Hospital
Locations (1):
- Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China